# Evaluating a Digital Peer Mentoring Platform With College Student Populations

NCT05764785

June 23, 2023



## INFORMED CONSENT FORM

University of Massachusetts Boston Department of Psychology 100 Morrissey Boulevard Boston, MA 02125-3393

Consent Form for "Evaluating the acceptability, feasibility, and efficacy of a digital peer mentoring platform with college student populations."

### **Introduction and Contact Information**

You are asked to take part in a research study. **Participation is voluntary.** The Principal Investigator is Dr. Jean Rhodes (Psychology Department, Faculty, UMass Boston). Please read this form and feel free to ask questions. If you have questions, Megyn Jasman will discuss them with you at <a href="maggyn.jasman001@umb.edu">megyn.jasman001@umb.edu</a>. The Principal Investigator can be reached at <a href="maggy-jean.rhodes@umb.edu">jean.rhodes@umb.edu</a>. The sponsor of the study is the National Institute of Mental Health.

## **Description of the Project:**

The purpose of the study is to assess the acceptability, feasibility, and efficacy of the MentorPRO application with the UMass Boston Directions for Student Potential (DSP) Summer Program.

We are seeking students who are members of one of Directions for Student Potential (DSP) Summer Program to complete 2 short virtual surveys (about 15-10 minutes each to complete) to help us evaluate the MentorPRO application (a technology platform for peer mentoring). If you decide to participate in this study, you will be asked to complete 2 short virtual surveys throughout the course of the project. 1 survey will be administered now (after this consent form, if you decide to participate), and the other will be 3 weeks after the end of the DSP Summer Program. All surveys will be administered virtually through Qualtrics links.

If you are eligible, you can receive \$50 for the first survey and \$50 for the final survey. Therefore, if you complete both surveys, you can earn up to \$100. Payment will be administered to participants via Tango Gift Cards at the end of the study.

If you agree to participate in the study and are eligible, you will be placed into 1 of 2 groups, based on your DSP cohort (a.m. or p.m. classes). One group of students will be asked to communicate with their mentor through MentorPRO (a technology platform for peer mentors that facilitates mentor-mentee communication and links mentees to third party mental health apps), while other students will be asked to communicate with their mentor as usual without MentorPRO.

The following data will also be requested from your academic records:

- Pre-matriculation/High school GPA
- Course load/credits for fall '23 semester

#### **Risks or Discomforts:**

The potential risks are minimal for this research project, as the procedures in this study that you will be exposed to are no more of a risk than what you encounter on a daily basis. You may experience some emotional discomfort related to assessment questions, which ask about academic performance, emotional wellbeing, and emotional and social functioning. If you wish to speak to someone further about these topics, you can reach UMass Boston's Counseling Center at <a href="mailto:counseling.center@umb.edu">counseling.center@umb.edu</a> or 617-287-5690.

You can skip any questions on the surveys that you would prefer not to answer, or you can stop participating at any time. This will not bear any negative consequences for you.

There is a risk for breach of confidentiality as participation in the research is dependent on membership in the DSP Program. We will do everything we can to protect your information. Some members from the research team will have access to identified data from the MentorPRO application (if in the MentorPRO group), from any third-party apps used through MentorPRO (if in the MentorPRO group), and surveys to match data across datasets. However, all analyses will be run on de-identified datasets and findings will be reported in aggregate form. We will do everything we can to protect your information.

## **Benefits:**

There is no direct benefit to you from participating in this study. Your participation may help us learn more about how to improve the integration of MentorPRO in college peer mentoring programs to best support students.

#### **Alternatives:**

Instead of being in this study, you can continue your current membership with the DSP program, and use of MentorPRO, without completing the study surveys.

#### **Confidentiality:**

Your participation in this research is **confidential**. That is, the information gathered for this project will not be published or presented in a way that would allow anyone to identify you. Information gathered for this project will be password protected and only the research team will have access to the data. However, if you are placed into the MentorPRO group, your mentor and DSP staff will have access to identified data on your engagement with any third-party apps you use. Only the research team, your mentor, and DSP staff will be able to see such engagement data. The Office for Human Research Protections (OHRP) in the U.S. Department of Health and Human Services (DHHS), the University of Massachusetts Boston Institutional Review Board (IRB) that oversees human research and other representatives of this organization may inspect and copy your information.

All data will be stored in password-protected folders. All identifiable information that could directly identify you (e.g., your name) will be removed from the datasets after the study has been completed. After we remove all identifiers, the information may also be used for future research or shared with other researchers without additional consent.

There are steps you can complete to protect your own privacy. For example, only taking the surveys in a private location without others around and closing out of your browser after taking the surveys will help maintain your privacy.

A description of this clinical trial will be available on http://www.clinicaltrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

There are no plans to share results of the study directly with participants.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena. There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations. Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

Please see below "Consent for Storing and Sharing of Data" for future storing and sharing of data.

#### Costs:

Participation in this study will be at no cost to you.

## **Voluntary Participation:**

The decision of whether or not to take part in this research study is voluntary. If you do decide to take part in this study, you may end your participation at any time without consequence. If you wish to end your participation, you should close out of the survey and the browser. If you would not like any of your data used for the study, please email Megyn Jasman (<a href="magyn.jasman001@umb.edu">megyn.jasman001@umb.edu</a>) to inform her that you wish for the researchers to not use your data for the purposes of the study. If you choose this, your survey data will be deleted.

Whatever you decide will in no way penalize you or involve a loss of benefits to which you are otherwise entitled. Choosing to not participate or stopping participation will not affect your standing with UMass Boston as a student, employee, etc, and will not affect your membership or participation in the DSP program or using MentorPRO. You can continue to use MentorPRO with your program as intended without participating (if you choose this, your data will not be used for the purposes of the research study). However, MentorPRO will continue to store your MentorPRO data.

There may be reasons for the PI to stop your participation in this study such as for administrative reasons or if the study is canceled. You will be told about any significant new information or changes in the study that could affect your willingness to continue participation.

## Other information:

The study PI, Jean Rhodes contributed seed funding toward the initial development of the MentorHub application, and the study PI turned over the company and all intellectual property to Academic Web Pages.

#### Questions:

If you have questions or if you have a research-related problem, Megyn Jasman will discuss them with you at <a href="megyn.jasman001@umb.edu">megyn.jasman001@umb.edu</a>. The Principal Investigator can be reached at <a href="jean.rhodes@umb.edu">jean.rhodes@umb.edu</a>.

If you have any questions or concerns about your rights as a research participant, please contact a representative of the Institutional Review Board (IRB), at the University of Massachusetts, Boston, which oversees research involving human participants. The Institutional Review Board may be reached by telephone or e-mail at (617) 287-5374 or at <a href="https://doi.org/numb.edu">https://doi.org/numb.edu</a>.

## Signatures:

I HAVE READ THE CONSENT FORM. MY QUESTIONS HAVE BEEN ANSWERED. CHECKING THE BELOW BOX MEANS THAT I CONSENT TO PARTICIPATE IN THIS STUDY.

By clicking the box, you are confirming that you are at least 18 years of age and are agreeing to participate in the research. You also agree to provide the research team with access to your pre-matriculation/high school GPA, as well as course load/credits for the Fall '23 semester. Please keep a copy of this form for your records or if you need to contact the research team.

# **Consent for Storing and Sharing of Data**

This study is collecting data from you. We would like to make your data is available for other research studies that may be done in the future. The research may be about similar or other types of research. These studies may be done by researchers at this institution or other institutions, including commercial entities. Our goal is to make more research possible. Identifiable data will be destroyed after the study is concluded.

Your data may be shared with researchers around the world. However, the decision to share your data is controlled by University of Massachusetts Boston. To get your data, future researchers must seek approval from University of Massachusetts Boston. The researchers must agree not to try to identify you.

We will do our best to protect your data during storage and when they are shared. However, there remains a possibility that someone could identify you. There is also the possibility that unauthorized people might access your data. In either case, we cannot reduce the risk to zero. You will not receive any direct benefit from sharing your data. However, sharing your data may contribute to research that could help others in the future. The use of your data may lead to new or other products or services with commercial value. These products or services could be patented and licensed. There are no plans to provide any payment to you should this occur.

Your name and identifying information will be removed from any data you provide before they are shared with other researchers. Researchers cannot easily link your identifying information to the data.

It is your choice whether or not to let researchers share your data for research in the future. If you say "yes," you can change your mind later. If you say "no," you can still fully participate in this study. If you change your mind

and no longer wish to have us store or share your data, you should contact Jean Rhodes, Ph.D. at 617-287-6368 or Jean.Rhodes@umb.edu. We will do our best to honor your request and to retrieve any data that has been shared with other researchers. However, there may be times we cannot. For example, if we do not have a way to identify your data we will not be able to retrieve them.

In addition, if the data have already been used for new research, the information from that research may still be used.

| Please indicate your choice: |
|-------------------------------------------------|
| YES, use my data in other research studies |
| NO, do NOT use my data in other research studie |